CLINICAL TRIAL: NCT07392385
Title: Effects of Volleyball-Specific Stroboscopic Training on Neuro-Psychophysiological Responses Across Different Experience Levels: A Randomized Controlled Trial
Brief Title: Neuro-Psychophysiological Characteristics of Athletes With Varying Levels of Experience
Acronym: NEPSY-SPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: The Scientific Research Project Fund of Yozgat Bozok University (Unknown)
Responsible Party: Principal Investigator, Izzet Kirkaya, Associate Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Bozok-SBF-IK-2025; 124C195 (Other: The Scientific Research Project Fund of Yozgat Bozok University (TÜBİTAK))
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Athletes; Sports Performance; Visual-Motor Processing; Neuro-Psychophysiological Responses in Athletes
Keywords: Stroboscopic Training; Dual-Task Performance; Functional Near-Infrared Spectroscopy; Electrodermal Activity; Eye Tracking; Athlete Experience Level

STUDY DESIGN:
Intervention Model Description: Participants will be stratified according to competitive experience level (novice, intermediate, and elite) and randomly assigned to either a stroboscopic training group or a control group using a parallel-group design. All participants will remain in their assigned study arm throughout the intervention period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to group allocation during data processing and analysis. Participants and care providers cannot be blinded due to the nature of the stroboscopic training intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroboscopic Training Group (Active Comparator): Participants will continue their regular volleyball training and perform the same volleyball-specific drills as the intervention group for 8 weeks. All exercises will be completed under normal visual conditions without the use of stroboscopic glasses.
  Interventions: Behavioral: Stroboscopic Volleyball Training
- Control Group (Active Comparator): Participants will continue their regular volleyball training and perform the same volleyball-specific drills as the intervention group for 8 weeks. All exercises will be completed under normal visual conditions without the use of stroboscopic glasses.
  Interventions: Behavioral: Conventional Volleyball Training (Control)

INTERVENTIONS:
Behavioral: Stroboscopic Volleyball Training — Participants will perform volleyball-specific training drills while wearing stroboscopic glasses that intermittently restrict visual input. The training will be conducted three times per week for 8 weeks, totaling 24 sessions. Each session will last approximately 35 minutes and will include volleyball-specific drills such as passing, setting, receiving, rotation-based movements, and reaction-based tasks. Visual disruption parameters of the stroboscopic glasses will be progressively adjusted throughout the intervention period.
  Arms: Stroboscopic Training Group
Behavioral: Conventional Volleyball Training (Control) — Participants will perform the same volleyball-specific training drills as the intervention group for 8 weeks under normal visual conditions, without the use of stroboscopic glasses. Training frequency, duration, and drill content will be matched to the intervention group.
  Arms: Control Group

SUMMARY:
This study aims to investigate the effects of an 8-week volleyball-specific stroboscopic training program on neuro-psychophysiological outcomes in female volleyball players with different levels of competitive experience. Participants will be categorized as novice, intermediate, or elite athletes and randomly assigned to either a stroboscopic training group or a control group. Both groups will continue their regular volleyball training, while only the intervention group will perform additional volleyball-specific drills using stroboscopic glasses. Neuro-psychophysiological assessments, including heart rate variability, electrodermal activity, functional near-infrared spectroscopy, dual-task performance, and eye-tracking measures, will be conducted before and after the training period. The study aims to determine whether stroboscopic training induces differential adaptations across experience levels and contributes to improved neuro-psychophysiological regulation associated with sport performance.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to examine the effects of volleyball-specific stroboscopic training on neuro-psychophysiological outcomes in athletes with different levels of competitive experience. Female volleyball players aged 10-16 years will be classified into three experience-based groups (novice, intermediate, and elite) according to their training history. Within each experience level, participants will be randomly assigned to either a stroboscopic training group or a control group, resulting in six study groups in total.

All participants will continue their routine volleyball training throughout the study period. In addition, athletes in the intervention group will complete an 8-week volleyball-specific stroboscopic training program, performed three times per week for a total of 24 sessions. Each training session will last approximately 35 minutes and will consist of volleyball-related drills, including passing, setting, receiving, rotation-based movements, and reaction-based tasks. Participants in the stroboscopic training group will perform these drills while wearing stroboscopic glasses with progressively adjusted visual disruption parameters, whereas the control group will perform the same drills under normal visual conditions.

Neuro-psychophysiological assessments will be conducted before and after the training period. Primary and secondary outcome measures will include heart rate variability, electrodermal activity, functional near-infrared spectroscopy recordings of prefrontal cortical activity, dual-task performance under varying levels of cognitive-motor demand, and eye-tracking parameters such as pupil diameter and fixation behavior. Psychological measures will also be collected using validated self-report instruments.

All measurements will be performed under standardized laboratory conditions. The study aims to determine whether stroboscopic training leads to differential neuro-psychophysiological adaptations across experience levels and whether such adaptations are associated with improved regulation of cognitive, physiological, and perceptual-motor processes relevant to volleyball performance.

ELIGIBILITY:
Inclusion Criteria:

* Female volleyball players aged 10 to 16 years
* Actively competing in organized volleyball
* Regular participation in team training sessions
* Classified as novice, intermediate, or elite based on training experience
* Written parental/legal guardian informed consent and participant assent obtained

Exclusion Criteria:

* Presence of any chronic medical condition affecting study outcomes
* Use of supplements or medications that may influence performance
* Current injury or participation in a rehabilitation program
* Failure to attend scheduled training sessions
* Inability to complete baseline or post-intervention assessments
* Injury occurring during the study period that prevents continued participation

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-06-21 (Actual)

PRIMARY OUTCOMES:
Prefrontal Cortical Activation (fNIRS) | Baseline (pre-intervention) and immediately after the 8-week intervention.
  Change in oxygenated and deoxygenated hemoglobin concentrations in the prefrontal cortex measured by functional near-infrared spectroscopy during dual-task performance
Heart Rate Variability (HRV) | Baseline (pre-intervention) and immediately after the 8-week intervention.
  Change in heart rate variability indices reflecting autonomic nervous system regulation, assessed at rest using a photoplethysmography-based system.
Dual-Task Performance | Baseline (pre-intervention) and immediately after the 8-week intervention.
  Change in reaction time and task performance under increasing levels of cognitive-motor demand assessed using a standardized dual-task protocol.
Electrodermal Activity (EDA) | Baseline (pre-intervention) and immediately after the 8-week intervention.
  Change in skin conductance responses reflecting sympathetic nervous system activity recorded during task performance.
Eye-Tracking Measures | Baseline (pre-intervention) and immediately after the 8-week intervention.
  Change in pupil diameter, fixation duration, and visual search behavior assessed using a wearable eye-tracking system during dual-task performance.

SECONDARY OUTCOMES:
Psychological Status (Depression, Anxiety, Stress) | Baseline (pre-intervention) and immediately after the 8-week intervention.
  Change in self-reported depression, anxiety, and stress levels assessed using a validated questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University Faculty of Sport Sciences, Yozgat, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Derived data only will be shared. No direct identifiers or sensitive personal information will be included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years thereafter.
Access Criteria: Access to de-identified individual participant data will be granted to qualified researchers upon reasonable request. Requests must include a brief research proposal and be approved by the study investigators to ensure consistency with the original ethical approval and data protection regulations. Data will be shared only for non-commercial research purposes and in accordance with institutional and legal requirements.

REFERENCES:
- [Background] Zhong X, Dai Y, Xu M, Jiang C. Volleyball training improves working memory in children aged 7 to 12 years old: an fNIRS study. Cereb Cortex. 2024 Jul 3;34(7):bhae275. doi: 10.1093/cercor/bhae275. PMID 39030744
- [Background] Zwierko M, Jedziniak W, Popowczak M, Rokita A. Effects of six-week stroboscopic training program on visuomotor reaction speed in goal-directed movements in young volleyball players: a study focusing on agility performance. BMC Sports Sci Med Rehabil. 2024 Feb 29;16(1):59. doi: 10.1186/s13102-024-00848-y. PMID 38424539
- [Background] Guo J, Zhao L, Liu G, Li H, Wu J. Stroboscopic training effects on athletic performance and cognitive function across populations, purposes, and skill types: a systematic review and meta-analysis of randomized controlled trials. Front Sports Act Living. 2025 Dec 11;7:1705693. doi: 10.3389/fspor.2025.1705693. eCollection 2025. PMID 41458106
- [Background] Piva T, Zerbini V, Barducco A, Mancioppi S, Raisi A, Vassali M, Bianchini G, Laporta M, Menegatti E, Grazzi G, Mazzoni G, Mandini S. Reduction in reaction time and improved oculomotor function following football-specific vision training in young players. BMC Sports Sci Med Rehabil. 2025 Oct 16;17(1):298. doi: 10.1186/s13102-025-01368-z. PMID 41102801
- [Background] Bherer L, Kramer AF, Peterson MS, Colcombe S, Erickson K, Becic E. Transfer effects in task-set cost and dual-task cost after dual-task training in older and younger adults: further evidence for cognitive plasticity in attentional control in late adulthood. Exp Aging Res. 2008 Jul-Sep;34(3):188-219. doi: 10.1080/03610730802070068. PMID 18568979
- [Background] Beavan A, Hanke L, Spielmann J, Skorski S, Mayer J, Meyer T, Fransen J. The effect of stroboscopic vision on performance in a football specific assessment. Sci Med Footb. 2021 Nov;5(4):317-322. doi: 10.1080/24733938.2020.1862420. Epub 2020 Dec 20. PMID 35077302